CLINICAL TRIAL: NCT04996732
Title: Studies on Long-term Survivorship of Discharged Patients With Malignant Tumor Based on Fudan University Shanghai Cancer Center Registry（FUCaRe）
Brief Title: Long-term Survivorship of Discharged Patients With Malignant Tumor Based on Single-institutional Cancer Registry
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ying Zheng, Director of Cancer Prevention Department, Fudan University Shanghai Cancer Center, Fudan University
Other Study IDs: YF-2021-01
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Neoplasms; Survival; Surgery; Radiotherapy; Drug Therapy
Keywords: Cancer; Survivorship
MeSH Terms: conditions — Neoplasms | interventions — Hospitalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Cancers: subgroups according to cancer sites
  Interventions: Procedure: hospitalization

INTERVENTIONS:
Procedure: hospitalization — Including various treatments such as surgery, radiotherapy, chemotherapy and immunotherapy during hospitalization

SUMMARY:
Real-world studies on long-term prognosis in patients who underwent anti-tumor treatments during hospitalization from a hospital-based cancer registry in china.

DETAILED DESCRIPTION:
This is a single-center continuous enrollment cohort study. The overall survival and disease-free survival of patients with malignant tumors in the target tumor hospital undergoing surgery, radiotherapy, chemotherapy, and immunotherapy were observed. Follow-up methods include medical records review, telephone call interview, and data linkage to the related provincial death certificate registries. This study will provide real world data-sets for researches on long-term survival and prognosis of cancer patients, and expend exploration on the cancer survival determinants both from clinical and social-economic prospective.

ELIGIBILITY:
Inclusion Criteria:

* All patients who completed tumor treatment (including surgery, radiotherapy, chemotherapy, immunotherapy, etc.) due to malignant tumors based on preoperative or intraoperative evaluation in Fudan University Shanghai Cancer Center during the study period.

Exclusion Criteria:

* Patients who have not been treated during hospitalization;
* Patients with non-malignant tumors.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who completed tumor treatment (including surgery, radiotherapy, chemotherapy, immunotherapy, etc.) due to malignant tumors based on preoperative or intraoperative evaluation in Fudan University Shanghai Cancer Center during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2041-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 15 years
  Death from any cause

SECONDARY OUTCOMES:
Disease-free survival | 15 years
  the time from treatment to recurrence of cancer, second primary cancer or death

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China